CLINICAL TRIAL: NCT04113850
Title: Mobile Acoustic Startle Reflex-monitoring System (MARS): A Pilot Study
Brief Title: Mobile Acoustic Startle Reflex-monitoring System (MARS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: School of Biomedical Sciences, University of Otago, Dunedin, New Zealand (Unknown); DigiTheronix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: IRB00217977
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single group, randomized (to sitting or standing postures)
Who Masked: Investigator
Masking Description: The study psychiatrist will be blind to MARS results at the time of the psychiatric interview that will confirm PTSD diagnosis and PTSD severity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting (Experimental): Subjects will undergo acoustic startle testing in the sitting position.
  Interventions: Device: Mobile Acoustic startle Reflex monitoring System (MARS)
- Standing (Experimental): Subjects will undergo acoustic startle testing in the standing position.
  Interventions: Device: Mobile Acoustic startle Reflex monitoring System (MARS)

INTERVENTIONS:
Device: Mobile Acoustic startle Reflex monitoring System (MARS) — Acoustic startle testing

SUMMARY:
This is a pilot study of 55 adult male veterans with PTSD. The study will test a new mobile application "app" that can be run on an iPhone10. The app, which is called the Mobile Acoustic startle Reflex-monitoring System (a.k.a., MARS), will be used to measure participant's acoustic startle in sitting or standing postures.

DETAILED DESCRIPTION:
The proposed study utilizes a randomized, controlled between-subjects design that will compare and contrast MARS data collected in the sitting versus standing position, and will determine the relationship between PTSD severity and MARS outcome measures. Fifty-five subjects will be recruited from Johns Hopkins and VA facilities, International Association of Fire Fighters Center of Excellence, Veteran Centers in Baltimore/District of Columbia/Northern Virginia area, as well as the Florida panhandle and through social media venues. When potential participants respond to advertisements, study coordinators will explain the purpose of the study and study procedures by phone before arranging a face-to-face meeting with the research team. Once a potential participant indicates willingness to participate, a study team member will meet with the participant at the their residence, or at the Johns Hopkins Bayview Medical Center, where the consent document will be reviewed and MARS testing will take place. Recruitment will continue until a total of 55 participants have been consented.

Volunteers shall sign a participation waiver acknowledging the inclusion/exclusion criteria and will be verbally briefed about the experimental proceedings. After consent procedures are complete, volunteers will provide a saliva sample and breathalyzer for "on the spot" drug screens. If drug screens are negative for sedatives and stimulants (both of which can alter the acoustic startle response), research volunteers will be interviewed using the Structured Interview for PTSD (SI-PTSD).

After completing the SI-PTSD (and it is clear that the subject meets criteria for PTSD), the subject will be be instructed to don earphones as well as noise insulating earmuffs. The MARS evaluation will then proceed in either a sitting or standing position, and the sound stimuli will be conducted at two frequencies [500 and 4000 Hertz (Hz)] at three volumes [65, 90, and 105 decibels (dBs)] for a total of 12 acoustic test sets, in random order. The MARS shall record both left and right eye reactions to each of these 12 acoustic/posture sets. The MARS protocol shall be administered for approximately 6 minutes while the volunteer is sitting/standing quietly and looking forward at the mobile device (which will be located approximately 60 centimeters away).

Within 3 weeks of MARS measurements, the study psychiatrist will conduct a private interview with the participant via remote video. The study psychiatrist (Dr. McCann), who will be blind to MARS data, will interview subjects using the Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual-5 (DSM-5) (CAPS-5).

Investigators will determine the statistical relationship between PTSD severity (as measured on a numerical scale from 1-5) and eye blink parameters. All data points will be entered into machine learning software (a.k.a. deep learning software) both to analyze interconnections between outcome measures and PTSD severity, but also to make predictions for future studies in PTSD patients evaluated using the MARS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PTSD

Exclusion Criteria:

* positive drug or alcohol screen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Acoustic Startle Response (speed) | 1 year after initiation of enrollment
  The acoustic startle response is the physiological measurement of eye-blink reflex following a sound. In the present protocol, various intensities of sound will be played using specialized equipment that plays sound through noise-cancelling earphones. The acoustic startle measure will be obtained using an "App" on an Apple iPhone 10. The primary startle response outcome is the time in seconds (typically milliseconds) between the playing of the sound, and the individual's eyeblink.

SECONDARY OUTCOMES:
Acoustic Startle Response (amplitude) | 1 year after the initiation of enrollment
  The acoustic startle response amplitude is a secondary outcome, and is defined as the maximal excursion of eye size from resting eye size, measured metrically (typically millimeters).

OTHER OUTCOMES:
Relationship between acoustic startle reflex and PTSD severity | 1 year after the initiation of enrollment
  The statistical correlation between acoustic startle response (both time and amplitude) and PTSD severity (as measured on a scale from 1 to 5) will be determined. In particular, individuals' average acoustic startle responses to each of the 12 stimuli parameters will be correlated with their PTSD severity. All 55 subjects will be included in these correlational analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Una McCann, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data analyses will be conducted by study investigators in New Zealand. Both sites (Baltimore and New Zealand) will have access to all study data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available to investigators in New Zealand at the time of data analyses, approximately one year after the study has begun.
Access Criteria: Only Dr. Yusuf Cakmak and data analyst (who will conduct the data analyses) will have access to the data. They will have a copy of the data which will be saved on a secure server.